CLINICAL TRIAL: NCT04305171
Title: Effect of Non-surgical Periodontal Treatment on Plasma Fibrinogen, Plasminogen Activator Inhibitor 1 and C-reactive Protein Levels in Cardiovascular Disease Patients With Periodontitis
Brief Title: Effect of Non-surgical Periodontal Treatment on Cardiovascular Risk Markers
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: MU-DT/PY-IRB 2018/022.0504
Record Dates: First submitted 2020-02-27; First posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Coronary Heart Disease; Periodontitis
Keywords: Coronary heart disease, peridontitis,
MeSH Terms: conditions — Coronary Disease; Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- coronary heart disease patients with periodontitis: Coronary heart disease patients confirmed through coronary angiography as having at least 50% diameter stenosis in at least one coronary artery and clinically stable with the absence of any potentially confounding inflammatory conditions for at least 6 months.
  Periodontitis classified as havingbleeding on probing (BOP), pocket depth (PD) > 4 mm, clinical attachment level (CAL) ≥ 5 mm and radiographic evidence of bone loss were presented at the same site of at least 4 teeth.
  Interventions: Procedure: non-surgical periodontal treatment
- coronary heart disease patients without periodontitisHD: Coronary heart disease patients confirmed through coronary angiography as having at least 50% diameter stenosis in at least one coronary artery and clinically stable with the absence of any potentially confounding inflammatory conditions for at least 6 months.
  Non-periodontitis classified as having PD ≤ 3 mm.
  Interventions: Procedure: non-surgical periodontal treatment
- non-coronary heart disease patients with periodontitis: Periodontitis classified as havingbleeding on probing (BOP), pocket depth (PD) > 4 mm, clinical attachment level (CAL) ≥ 5 mm and radiographic evidence of bone loss were presented at the same site of at least 4 teeth.
  Interventions: Procedure: non-surgical periodontal treatment
- non-coronary heart disease patients without periodontitis: Non-periodontitis classified as having PD ≤ 3 mm.
  Interventions: Procedure: non-surgical periodontal treatment

INTERVENTIONS:
Procedure: non-surgical periodontal treatment — scaling and root planing, home care instruction

SUMMARY:
The research question was to investigate whether non-surgical periodontal therapy could reduce cardiovascular risk markers in Coronary heart disease (CHD) patients.

DETAILED DESCRIPTION:
CHD patients or non-CHD with or without periodontitis were included. They were provided with non-surgical periodontal therapy (NSPT). Periodontal parameters and cardiovascular risk markers were measured at baseline and 3 months and 6 months after NSPT.

ELIGIBILITY:
Inclusion Criteria:

* non-CHD or CHD (at least 50% diameter stenosis in at least one coronary artery and clinically stable with absence of any potentially confounding inflammatory conditions for at least 6 months)
* had at least 14 natural teeth excluding third molars

Exclusion Criteria:

* received anticoagulant drugs
* had chronic conditions (e.g. diabetes mellitus, rheumatoid arthritis, malignancy, autoimmune disease) or acute conditions (e.g. trauma, surgery) or medications known to affect systemic inflammatory markers (e.g. antibiotics, immunosuppressive, contraceptives) within 3 months
* pregnancy or lactation
* presence or history of other infections
* periodontal treatment within 6 months
* tooth extractions within 2 months prior to the study.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatients who came to the Hospital for Tropical Medicine, Faculty of Tropical Medicine, Mahidol University or Rajavithi Hospital, Thailand
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
change in fibrinogen level between baseline and 3 months after non-surgical periodontal treatment | 3 months after non-surgical periodontal treatment
  change in plasma fibrinogen level (pg/mL)
change in activator inhibitor 1 between baseline and 3 months after non-surgical periodontal treatment | 3 months after non-surgical periodontal treatment
  change in activator inhibitor 1 level (pg/mL)
change in C-reactive protein between baseline and 3 months after non-surgical periodontal treatment | 3 months after non-surgical periodontal treatment
  change in C-reactive protein level (mg/L)
change in fibrinogen level between baseline and 6 months after non-surgical periodontal treatment | 6 months after non-surgical periodontal treatment
  change in plasma fibrinogen level (pg/mL)
change in activator inhibitor 1 between baseline and 6 months after non-surgical periodontal treatment | 6 months after non-surgical periodontal treatment
  change in activator inhibitor 1 level (pg/mL)
change in C-reactive protein between baseline and 6 months after non-surgical periodontal treatment | 6 months after non-surgical periodontal treatment
  change in C-reactive protein level (mg/L)

SECONDARY OUTCOMES:
change of bleeding on probing between baseline and 3 months after non-surgical periodontal treatment | 3 months after non-surgical periodontal treatment
  percetage of sites with bleeding on probing
change of pocket depth between baseline and 3 months after non-surgical periodontal treatment | 3 months after non-surgical periodontal treatment
  Depth of periodontal pocket in millimeters
change of clinical attachment level between baseline and 3 months after non-surgical periodontal treatment | 3 months after non-surgical periodontal treatment
  Level of clinical attachment in millimeters
change of bleeding on probing between baseline and 6 months after non-surgical periodontal treatment | 6 months after non-surgical periodontal treatment
  percetage of sites with bleeding on probing
change of pocket depth between baseline and 6 months after non-surgical periodontal treatment | 6 months after non-surgical periodontal treatment
  Depth of periodontal pocket in millimeters
change of clinical attachment level between baseline and 6 months after non-surgical periodontal treatment | 6 months after non-surgical periodontal treatment
  Level of clinical attachment in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Supanee Rassameemasmaung, PhD, Principal Investigator — Mahidol University Faculty of Dentistry
Locations (3):
- Thailand (3):
  - Department of Clinical Tropical Medicine, Faculty of Tropical Medicine, Mahidol University, Ratchathewi, Bangkok
  - Department of Medicine, Rajavithi Hospital, Ratchathewi, Bangkok
  - Mahidol University Faculty of Dentistry, Ratchathewi, Bangkok

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ye Z, Cao Y, Miao C, Liu W, Dong L, Lv Z, Iheozor-Ejiofor Z, Li C. Periodontal therapy for primary or secondary prevention of cardiovascular disease in people with periodontitis. Cochrane Database Syst Rev. 2022 Oct 4;10(10):CD009197. doi: 10.1002/14651858.CD009197.pub5. PMID 36194420